CLINICAL TRIAL: NCT05362279
Title: The Effect of Training on Oxygen Therapy With High Flow Nasal Cannula on the Knowledge Level of Pediatric Nurses; A Randomized Controlled Trial
Brief Title: The Effect of Education on Nurses' Knowledge About High-flow Nasal Cannula Oxygen Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Aslı Alaca, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAlaca
Record Dates: First submitted 2022-04-23; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Pediatric
Keywords: HFNC; Nursing Care; Knowledge Level; Education

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with pretest-posttest experimental and control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test after post-test training (Experimental): Pre-test will be applied to the nurses in the experimental group before the training. The post-test will be applied to the experimental group, to which the pre-test was applied, one month after the training was given.
  Interventions: Other: Training
- Test without training (No Intervention): The nurses in the control group are the group to be administered the post-test without any intervention after the pre-test. The post-test will be administered one month after the pre-test.

INTERVENTIONS:
Other: Training — One month after the pre-test, the post-test will be administered to the nurses who will be in the control group.
  Nurses who will be in the experimental group will be given training after the pre-test. A post-test will be administered one month after the training.
  Arms: Test after post-test training

SUMMARY:
This study was conducted to evaluate the oxygen therapy methods used in pediatric services and to specify the roles and responsibilities of nurses in the application of HFNC, which is one of these methods. Although the decision to implement this treatment method is under the responsibility of the physician in Turkey, the use of the device, observing the effectiveness of the treatment, monitoring and recording the changes in the vital signs of the children are under the responsibility of the nurses shows the importance of the nursing perspective on HFNC.

DETAILED DESCRIPTION:
High-flow nasal cannula oxygen therapy (HFNC) which meets the patient's ventilation need is a non-invasive ventilation system in which warmed and humidified oxygen is administered to the patient at varying flows with the help of a nasal cannula.This study will be conducted as a randomized controlled study with the participation of 70 nurses working in the pediatric clinics of a public hospital between December 2021 and May 2022, as an experimental group (n=35) and a control group (n=35). In the study, two-stage sampling method will be used to determine the nurses who will take place in the experimental and control groups. After the nurses are stratified according to their professional years, assignment to the experimental and control groups will be made by simple random sampling method. The experimental group will be given a pre-test before the training and a post-test one month after the training. In order to avoid interaction between the two groups, the data of the nurses in the control group will be collected first. The knowledge level of the nurses in the experimental and control groups will be evaluated with the HFNC Information Form.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in any of the pediatric emergency departments, pediatric clinics
* No previous training in HFNC treatment
* Follow-up of patients treated with HFNC
* Volunteering to participate in research

Exclusion Criteria:

* Those who have received in-service training on HFNC implementation
* Those who work as responsible nurses or training nurses in the clinics where the research will be conducted

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-05-10 (Estimated); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Knowledge Level - Education Form- Questionnaire | One month after training
  To increase the knowledge level of nurses about oxygen therapy with high flow nasal cannula.

CONTACTS AND LOCATIONS:
Overall Officials: Aslı ALACA, Principal Investigator — Study Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colleti Junior J, Longui TE, Carvalho WB. HIGH-FLOW NASAL CANNULA POST-TRACHEAL EXTUBATION IN A CHILD WITH UPPER AIRWAY OBSTRUCTION: CASE REPORT. Rev Paul Pediatr. 2018 Jul-Sep;36(3):372-375. doi: 10.1590/1984-0462/;2018;36;3;00010. Epub 2018 Jul 10. PMID 29995143